CLINICAL TRIAL: NCT01073020
Title: Surgery or Lifestyle With Intensive Medical Management in the Treatment of Type 2 Diabetes (SLIMM-T2D)
Brief Title: Surgery or Lifestyle With Intensive Medical Management in the Treatment of Type 2 Diabetes
Acronym: SLIMM-T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009P-001610
Record Dates: First submitted 2010-02-16; First posted 2010-02-22 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Type 2 Diabetes Mellitus; Obesity; Lifestyle; Bariatric Surgery; Laparoscopic Adjustable Gastric Band; Laparoscopic Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Gastric Bypass; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Gastric Band vs Intensive Diabetes & Weight Management (Active Comparator): Patients will be randomized to receive either 1) laparoscopic placement of an adjustable gastric band (LAGB) or 2) treatment with an intensive medical and weight management (IMWM) program.
  LAGB will be placed using the "pars flaccida" technique. The Allergan laparoscopic band "LAP BAND" system will be utilized. LAGB ports will be placed in subcutaneous pockets in the right upper abdomen.
  The IMWM group will participate in the Weight Achievement and Intensive Treatment (Why WAIT) program, which is a multidisciplinary program for weight control and intensive diabetes management designed by Joslin Diabetes Center. Key aspects include: 1) Intensive and interactive medication adjustments, 2) Structured modified dietary intervention, 3) Graded, balanced, and individualized exercise intervention, 4) Cognitive behavioral intervention and 5) Group education.
  Interventions: Device: Allergan Adjustable Gastric Band Surgery; Other: Intensive Medical Diabetes & Weight Management (Why WAIT) - Band Group
- RYGB vs Intensive Diabetes & Weight Management (Active Comparator): Patients will be randomized to receive either 1) Roux-en-Y gastric bypass (RYGB) surgery or 2) treatment with an intensive medical and weight management (IMWM) program.
  RYGB will be performed using a 75 cm antecolic, ante-gastric Roux limb created with a 50 cm pancreaticobiliary limb. A 15-20 cc gastric pouch will be created lying along the lesser curve of the stomach, with division of the vagal trunks at the lower border of the pouch.
  The IMWM group will participate in the Weight Achievement and Intensive Treatment (Why WAIT) program, which is a multidisciplinary program for weight control and intensive diabetes management designed by Joslin Diabetes Center. Key aspects include: 1) Intensive and interactive medication adjustments, 2) Structured modified dietary intervention, 3) Graded, balanced, and individualized exercise intervention, 4) Cognitive behavioral intervention and 5) Group education.
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGB) Surgery; Other: Intensive Medical Diabetes & Weight Management (Why WAIT) - Bypass Group

INTERVENTIONS:
Device: Allergan Adjustable Gastric Band Surgery
  Arms: Gastric Band vs Intensive Diabetes & Weight Management
Other: Intensive Medical Diabetes & Weight Management (Why WAIT) - Band Group — Intensive Medical Diabetes & Weight Management (Why WAIT) - Band Group
  Arms: Gastric Band vs Intensive Diabetes & Weight Management
Procedure: Roux-en-Y Gastric Bypass (RYGB) Surgery
  Arms: RYGB vs Intensive Diabetes & Weight Management
Other: Intensive Medical Diabetes & Weight Management (Why WAIT) - Bypass Group — Intensive Medical Diabetes & Weight Management (Why WAIT) - Bypass Group
  Arms: RYGB vs Intensive Diabetes & Weight Management

SUMMARY:
There is substantial clinical evidence regarding the safety and efficacy of currently practiced bariatric surgical techniques to improve metabolic control and/or resolve type 2 diabetes (T2DM) in clinically severe obese patients (class 3 obesity). Evidence suggests such procedures have greater effects on insulin secretion and insulin action than that expected from weight loss alone, which has led to the recent claim that such procedures may be useful as a primary treatment for T2DM in the moderately obese population. Concurrently, there have also been substantial advances in the non-surgical medical management of T2DM. As a result, the best treatment algorithm for T2DM patients with class 1 & 2 obesity is increasingly controversial. This trial investigates the utility of currently practiced and available bariatric surgical procedures as compared with multidisciplinary intensive medical and weight management for the treatment of T2DM with class 1 and 2 obesity.

DETAILED DESCRIPTION:
Primary Specific Aim 1: To evaluate the effectiveness of laparoscopic adjustable gastric band versus intensive medical and weight management in the treatment of T2DM.

There has been only one randomized control trial to date comparing surgical to medical management of T2DM in the less obese population, which demonstrated substantial superiority of the laparoscopic adjustable gastric band (LAGB) in the improvement of glycemic and metabolic measures. However, these findings remain controversial as the magnitude of weight loss in this study was far superior to that generally reported following LAGB. Thus, we propose a second prospective randomized trial to evaluate the effectiveness of intensive medical and weight management (IMWM) vs. LAGB in T2DM patients with BMI in the 30-42 kg/m^2 range. This range does extend LAGB surgery to BMI limits below those currently used in medical care, FDA Investigational Device Exemption (IDE) G090163. The primary outcome variable will be attaining glycemic control (as defined by fasting plasma glucose levels <126 mg/dL and HbA1c <6.5%) at one year of follow-up. The study was subsequently extended to 3 years, with the same outcome measures.

Primary Specific Aim 2: To evaluate the effectiveness of laparoscopic Roux-en-Y gastric bypass versus intensive medical and weight management in the treatment of T2DM.

Although observational studies and meta-analyses suggest rapid and sustained improvement or resolution of diabetes following laparoscopic Roux-en-Y gastric bypass (LRYGB), to date there has been no randomized trial directly comparing these effects to those produced by IMWM. We propose a prospective randomized trial comparing the effectiveness of IMWM vs. LRYGB in T2DM patients with BMI's in the 30-42 kg/m^2 range. This range extends LRYGB surgery to BMI limits below those currently used in medical care to explore the use of this type of surgical procedure in type 2 diabetes with lesser magnitude obesity. The primary outcome variable will be attaining glycemic control (as defined by fasting plasma glucose levels <126 mg/dL and HbA1c <6.5%) at one year of follow-up. The study was subsequently extended to 3 years, with the same outcome measures.

The trial is designed to allow for strong patient preference towards specific surgical procedures, and as such is designed as two parallel trials with each of the two surgical procedures judged against intensive medical weight management. Subjects without strong preference will be randomly assigned to one of the four study arms.

Secondary Specific Aims:

Determination of suitable study design: In addition to testing the effectiveness of current and available surgical techniques as compared to medical management, this trial will also test the utility of this trial design in future multi-institutional comparative effectiveness studies of these therapies, or alternatively, in future trials evaluating new surgical procedures being designed specifically for less obese T2DM patients.

Measurement of metabolic factors: Insulin secretion and action will be assessed during provocative mixed meal tolerance tests (MMTT) using the corrected incremental insulin response (CIR) and the composite insulin sensitivity index (CISI). MMTT will be performed in all groups at baseline and repeated at the time point of 10% weight loss (matched for weight loss), and at 12 months following randomization (matched for time).

Measurement of cardiovascular risk factors: Each group will be studied for evidence of changes in cardiovascular disease risk factors. Multiple surrogate measures of cardiovascular health will be compared, including blood pressure, fasting lipid profiles, endothelium-dependent vasodilatation and plasma will be collected for circulating markers of endothelial function. The study was subsequently extended to 3 years, with the same outcome measures.

Measurement of metabolic rate: Each group will be studied for change in energy expenditure and respiratory quotient using the non-invasive indirect calorimetry technique.

Quality of life and cost utility outcomes: Longitudinal measures of patient reported quality of life outcomes, and cost utility measures will also be collected to generate preliminary data for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be those with T2DM, with a diagnosis of diabetes of at least one year in duration,
* BMI 30-45 kg/m^2 for the LAGB compared to intensive medical weight and diabetes management and BMI 30-42 kg/m^2 for LRYGB compared to intensive medical weight and diabetes management,
* Age 21-65 years,
* With a strong desire for substantial weight loss, who are free from active cardiovascular or other diseases that would render them unable to partake in a structured exercise program or to undergo a bariatric surgical procedure, and who are committed to life long medical and nutritional follow up.

Exclusion Criteria:

* Detectable levels of glutamic acid decarboxylase (GAD) antibody or a history of diabetic ketoacidosis or uncontrolled T2DM (consistent fasting blood glucose >200 mg/dl or HbA1c above twice normal);
* Previous gastrointestinal surgery, inflammatory bowel disease, esophageal diseases including severe intractable esophagitis, Barrett's Disease, esophageal dysmotility or other impaired gastric motility (gastroparesis), or hiatal hernia >3 cm in size, chronic or acute bleeding conditions including peptic ulcer disease, portal hypertension (gastric or esophageal varices), chronic pancreatitis, or cirrhosis of the liver;
* Malignant or debilitating medical conditions, severe cardiopulmonary disease including uncontrolled hypertension (repeated systolic measures >160 or diastolic > 95 mm Hg on more than one day), unstable angina pectoris, recent myocardial infarction within 6 months, history of coronary artery bypass surgery or angioplasty, congestive heart failure, arrhythmia, stroke or transient ischemic attacks, urinary albumin excretion >300 mcg/mg creatinine and/or serum creatinine >1.5 mg/dL (permitting safety of increased dietary protein intake),
* Any endocrine disorder other than T2DM or thyroid disease which is stable on replacement therapy, including Cushing's syndrome;
* Any previous history of eating disorders, history of drug and/or alcohol abuse within 2 years of the screening visit, history of impaired mental status as defined by Diagnostic and Statistical Manual, 4th Edition (DSM-4) criteria and including, but not limited to active substance abuse, a history of schizophrenia, borderline personality disorder, uncontrolled depression, suicidal attempts within the past two years or current suicidal tendencies or ideations.
* Subjects will be excluded if there is a history of significant weight loss (>3%) within the previous 3 months or participation in alternate medically supervised exercise or weight reduction program within the previous 3 months, or with use of prescription or over the counter weight reduction medications or supplements within one month of the Screening Visit and for the duration of study participation.
* Women who are lactating, planning pregnancy, or unwilling to use contraception during the course of the trial.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison B. Goldfine, MD, Principal Investigator — Joslin Diabetes Center; Ashley Vernon, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lautz D, Halperin F, Goebel-Fabbri A, Goldfine AB. The great debate: medicine or surgery: what is best for the patient with type 2 diabetes? Diabetes Care. 2011 Mar;34(3):763-70. doi: 10.2337/dc10-1859. No abstract available. PMID 21357363
- [Result] Halperin F, Ding SA, Simonson DC, Panosian J, Goebel-Fabbri A, Wewalka M, Hamdy O, Abrahamson M, Clancy K, Foster K, Lautz D, Vernon A, Goldfine AB. Roux-en-Y gastric bypass surgery or lifestyle with intensive medical management in patients with type 2 diabetes: feasibility and 1-year results of a randomized clinical trial. JAMA Surg. 2014 Jul;149(7):716-26. doi: 10.1001/jamasurg.2014.514. PMID 24899464
- [Result] Ding SA, Simonson DC, Wewalka M, Halperin F, Foster K, Goebel-Fabbri A, Hamdy O, Clancy K, Lautz D, Vernon A, Goldfine AB. Adjustable Gastric Band Surgery or Medical Management in Patients With Type 2 Diabetes: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2015 Jul;100(7):2546-56. doi: 10.1210/jc.2015-1443. Epub 2015 Apr 24. PMID 25909333
- [Result] Yu EW, Wewalka M, Ding SA, Simonson DC, Foster K, Holst JJ, Vernon A, Goldfine AB, Halperin F. Effects of Gastric Bypass and Gastric Banding on Bone Remodeling in Obese Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2016 Feb;101(2):714-22. doi: 10.1210/jc.2015-3437. Epub 2015 Nov 24. PMID 26600045
- [Result] Panosian J, Ding SA, Wewalka M, Simonson DC, Goebel-Fabbri A, Foster K, Halperin F, Vernon A, Goldfine AB. Physical Activity in Obese Type 2 Diabetes After Gastric Bypass or Medical Management. Am J Med. 2017 Jan;130(1):83-92. doi: 10.1016/j.amjmed.2016.07.019. Epub 2016 Aug 20. PMID 27555097
- [Result] Simonson DC, Halperin F, Foster K, Vernon A, Goldfine AB. Clinical and Patient-Centered Outcomes in Obese Patients With Type 2 Diabetes 3 Years After Randomization to Roux-en-Y Gastric Bypass Surgery Versus Intensive Lifestyle Management: The SLIMM-T2D Study. Diabetes Care. 2018 Apr;41(4):670-679. doi: 10.2337/dc17-0487. Epub 2018 Feb 6. PMID 29432125
- [Result] Simonson DC, Vernon A, Foster K, Halperin F, Patti ME, Goldfine AB. Adjustable gastric band surgery or medical management in patients with type 2 diabetes and obesity: three-year results of a randomized trial. Surg Obes Relat Dis. 2019 Dec;15(12):2052-2059. doi: 10.1016/j.soard.2019.03.038. Epub 2019 Apr 16. PMID 31931977
- [Derived] Dreyfuss JM, Yuchi Y, Dong X, Efthymiou V, Pan H, Simonson DC, Vernon A, Halperin F, Aryal P, Konkar A, Sebastian Y, Higgs BW, Grimsby J, Rondinone CM, Kasif S, Kahn BB, Foster K, Seeley R, Goldfine A, Djordjilovic V, Patti ME. High-throughput mediation analysis of human proteome and metabolome identifies mediators of post-bariatric surgical diabetes control. Nat Commun. 2021 Nov 29;12(1):6951. doi: 10.1038/s41467-021-27289-2. PMID 34845204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be recruited from the Joslin Diabetes Center and Partners Healthcare. All patients with type 2 diabetes (T2DM) attending the Brigham and Women's Hospital (BWH) Bariatric Surgery Program orientation sessions (>1200 subjects/year) will be presented with this trial as an option. Recruitment will also be from the >13,000 T2DM patients who receive their medical care at Joslin Diabetes Center or the Partners Healthcare Primary Care Network.
Pre-assignment Details: After initial contact, patients will undergo the following: 1) Telephone screening (review inclusion and exclusion criteria, description of interventions), 2) Attend clinical trial orientation session (detailed description of interventions, protocol, procedures, surgical clearance, nutritional evaluation, risks, benefits), 3) Medical and surgical screening visit (sign informed consent, screening lab tests, history and physical, psychological evaluation for bariatric surgery, exercise clearance).
Groups:
- Laparoscopic Adjustable Gastric Band (LAGB): Laparoscopic Adjustable Gastric Band (LAGB): Allergan Adjustable Gastric Band (Device)
  Participants were randomized to LAGB vs. an intensive medical diabetes and weight management program (Why Wait? Program)
- Intensive Medical Diabetes & Weight Management (LAGB Grp): Participants were randomized to LAGB vs. an intensive medical diabetes and weight management program (Why Wait? Program)
- RYGB: Roux-en-Y Gastric Bypass (Surgery)
  Participants were randomized to RYGB vs. an intensive medical diabetes and weight management program (Why WAIT? Program)
- Intensive Medical Diabetes & Weight Management (RYGB Grp): Participants were randomized to RYGB vs. an intensive medical diabetes and weight management program (Why Wait? Program)
Period: Overall Study
Arm/Group | Laparoscopic Adjustable Gastric Band (LAGB) | Intensive Medical Diabetes & Weight Management (LAGB Grp) | RYGB | Intensive Medical Diabetes & Weight Management (RYGB Grp)
Started | 23 | 22 | 22 | 21
Completed | 16 | 17 | 19 | 19
Not Completed | 7 | 5 | 3 | 2
Not completed — Withdrawal by Subject | 6 | 4 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 2 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants first selected whether they preferred gastric band or RYGB. After consent, they were randomized to either surgery or intensive medical diabetes and weight management. This resulted in 2 independent substudies, one of which compared band to its corresponding intensive medical diabetes and weight management group, and one of which compared RYGB to its corresponding intensive medical diabetes and weight management group..
Groups:
- Laparoscopic Adjustable Gastric Band (LAGB): Laparoscopic Adjustable Gastric Band: Allergan Adjustable Gastric Band (Device)
- Intensive Medical Diabetes & Weight Management (LAGB Group): Intensive Medical Diabetes & Weight Management: Intensive Medical Diabetes & Weight Management (LAGB Group)
  This group selected band as preferred surgery, but were randomized to medical management.
- RYGB: Roux-en-Y Gastric Bypass (Surgery)
- Intnnsive Medical Diabetes and Weight Management (RYGB Group): Intensive Medical Diabetes & Weight Management: Intensive Medical Diabetes & Weight Management (RYGB Group)
  This group selected RYGB as preferred surgery, but were randomized to medical management.
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Adjustable Gastric Band (LAGB) | Intensive Medical Diabetes & Weight Management (LAGB Group) | RYGB | Intnnsive Medical Diabetes and Weight Management (RYGB Group) | Total
Number analyzed (Participants) | 23 | 22 | 22 | 21 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 22 | 21 | 88
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (12.1) | 51.4 (7.5) | 50.7 (7.6) | 52.6 (4.3) | 51.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 16 | 10 | 47
  Male | 11 | 13 | 6 | 11 | 41
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 22 | 21 | 88

OUTCOME MEASURES:

1. Primary Outcome: Fasting Plasma Glucose <126 mg/dL and HbA1c < 6.5% at Three Years of Follow-up.
Description: The primary outcome variable of both parallel trials will be the percent of patients attaining glycemic control (defined as fasting plasma glucose < 126 mg/dL and HbA1c < 6.5%) at three years of follow-up.
Time Frame: 3 years
Population: Patients not analyzed include: 7 of 23 in LAGB (4 withdrew consent before intervention,1 determined to not be a surgical candidate before intervention, and 2 withdrew consent between 1 and 3 years); 5 of 22 in IMWM (LAGB Grp) (4 withdrew consent, 1 death); 3 of 22 in the RYGB group (1 withdrew consent; 1 breast cancer diagnosis and 1 psychiatric illness pre-intervention); 2 of 21 IMWM (RYGB Grp) withdrew consent before intervention.
Measure: Number; unit: % of patients
Groups:
- LAGB: Laparoscopic Adjustable Gastric Band: Allergan Adjustable Gastric Band (Device)
  Participants were randomized to LAGB vs. an intensive medical diabetes and weight management program (Why WAIT? Program)
Arm/Group | LAGB | Intensive Medical Diabetes & Weight Management (LAGB Grp) | RYGB | Intensive Medical Diabetes & Weight Management (RYGB Grp)
Number analyzed (Participants) | 16 | 17 | 19 | 19
% of patients | 13 | 5 | 42 | 0
Statistical Analysis 1: Comparison: LAGB vs Intensive Medical Diabetes & Weight Management (LAGB Grp); Test type: Superiority; p = 0.60, Chi-squared; proportion = 0.08 — Estimation parameter is the difference between the proportion of patients in the LAGB group vs. proportion of patients in the Intensive Medical Diabetes & Weight Management (LAGB Grp) who achieved the primary outcome
Statistical Analysis 2: Comparison: RYGB vs Intensive Medical Diabetes & Weight Management (RYGB Grp); Test type: Superiority; p = 0.005, Chi-squared; proportion = 0.42 — Estimation parameter is the difference between the proportion of patients in the RYGB group vs. proportion of patients in the Intensive Medical Diabetes & Weight Management (RYGB Grp) who achieved the primary outcome

2. Secondary Outcome: Glycemic Control, as Measured by Hemoglobin A1c
Description: All participants had type 2 diabetes. Long-term diabetes control is typically evaluated in both clinical and research settings using the measurement of Hemoglobin A1c (a measure of glycated hemoglobin, proportional to average glucose levels over approximately 3 months). This endpoint (hemoglobin A1c) was measured at 3 years after intervention. Reported values are changes from baseline derived from the mixed effects model analysis, adjusted for baseline.
Time Frame: 3 years
Population: Randomized patients who had at least one post-randomization visit (modified intention to treat).
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | LAGB | Intensive Medical Diabetes & Weight Management (LAGB Grp) | RYGB | Intensive Medical Diabetes & Weight Management (RYGB Grp)
Number analyzed (Participants) | 16 | 17 | 19 | 19
Percent | -0.8 [-1.6 to -0.0] | 0.2 [-0.6 to 1.0] | -1.8 [-2.4 to -1.2] | -0.4 [-1.1 to 0.3]
Statistical Analysis 1: Comparison: LAGB vs Intensive Medical Diabetes & Weight Management (LAGB Grp); Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Net) = 1.0 — Estimation parameter is the difference between the change from baseline in HbA1c in the LAGB group vs. change from baseline in HbA1c in the Intensive Medical Diabetes & Weight Management (LAGB Grp), adjusted for baseline HbA1c
Statistical Analysis 2: Comparison: RYGB vs Intensive Medical Diabetes & Weight Management (RYGB Grp); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.4 — Estimation parameter is the difference between the change from baseline in HbA1c in the RYGB group vs. change from baseline in HbA1c in the Intensive Medical Diabetes & Weight Management (RYGB Grp), adjusted for baseline HbA1c

3. Secondary Outcome: Body Mass Index
Description: Change in body mass index 3 years after intervention
Time Frame: 3 years
Population: Randomized patients who had at least one post-randomization visit (modified intention to treat).
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | LAGB | Intensive Medical Diabetes & Weight Management (LAGB Grp) | RYGB | Intensive Medical Diabetes & Weight Management (RYGB Grp)
Number analyzed (Participants) | 16 | 17 | 19 | 19
kg/m^2 | -3.9 [-5.2 to -2.6] | -1.7 [-3.0 to 0.4] | -8.7 [-10.3 to -7.1] | -4.1 [-8.8 to 0.6]
Statistical Analysis 1: Comparison: LAGB vs Intensive Medical Diabetes & Weight Management (LAGB Grp); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 2.2 — Estimation parameter is the difference between the change from baseline in BMI in the LAGB group vs. change from baseline in BMI in the Intensive Medical Diabetes & Weight Management (LAGB Grp), adjusted for baseline BMI
Statistical Analysis 2: Comparison: RYGB vs Intensive Medical Diabetes & Weight Management (RYGB Grp); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 4.6 — Estimation parameter is the difference between the change from baseline in BMI in the RYGB group vs. change from baseline in BMI in the Intensive Medical Diabetes & Weight Management (RYGB Grp), adjusted for baseline BMI

4. Secondary Outcome: Cardiovascular Risk
Description: UKPDS risk of coronary heart disease, reported as change from baseline
Time Frame: 3 years
Population: Patients who had at least one post-randomization visit were analyzed (modified intention to treat).
Measure: Mean (95% Confidence Interval); unit: percent likelihood of event in next 10 y
Arm/Group | LAGB | Intensive Medical Diabetes & Weight Management (LAGB Grp) | RYGB | Intensive Medical Diabetes & Weight Management (RYGB Grp)
Number analyzed (Participants) | 16 | 17 | 19 | 19
percent likelihood of event in next 10 y | 0.7 [-1.4 to 2.8] | 2.2 [0.2 to 4.2] | -2.5 [-4.3 to -0.7] | 0.1 [-2.0 to 2.1]
Statistical Analysis 1: Comparison: LAGB vs Intensive Medical Diabetes & Weight Management (LAGB Grp) vs RYGB vs Intensive Medical Diabetes & Weight Management (RYGB Grp); Test type: Superiority; p = 0.81, Mixed Models Analysis; Mean Difference (Net) = 1.5 — Estimation parameter is the difference between change from baseline in CHD risk over 10 yrs. in LAGB group vs. change from baseline in CHD risk over 10 yrs. in Intensive Medical Diabetes & Weight Management (LAGB Grp), adjusted for baseline CHD risk
Statistical Analysis 2: Comparison: RYGB vs Intensive Medical Diabetes & Weight Management (RYGB Grp); Test type: Superiority; p = 0.009, Mixed Models Analysis; Mean Difference (Net) = 2.6 — Estimation parameter is the difference between change from baseline in CHD risk over 10 yrs. in RYGB group vs. change from baseline in CHD risk over 10 yrs. in Intensive Medical Diabetes & Weight Management (RYGB Grp), adjusted for baseline CHD risk

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events (AE), including all-cause mortality, serious, and other adverse events were monitored in all participants, and information is included in this report. For those who were lost to followup, AE were recorded up to the timepoint of loss to followup. The total number of participants indicated is the number who completed 3 years of followup, and thus for whom AE monitoring was complete for the 3 year study.
Groups:
- Laparoscopic Adjustable Gastric Band Surgery: Surgical Implantation of Allergan Adjustable Gastric Band (Device)
Arm/Group | Laparoscopic Adjustable Gastric Band Surgery | Intensive Medical Diabetes and Weight Management: Band Group | Roux-en-Y Gastric Bypass (RYGB) Surgery | Intensive Medical Diabetes and Weight Management: RYGB Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/22 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 9/18 | 6/22 | 11/19 | 5/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22 | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Adjustable Gastric Band Surgery (N=18) | Intensive Medical Diabetes and Weight Management: Band Group (N=22) | Roux-en-Y Gastric Bypass (RYGB) Surgery (N=19) | Intensive Medical Diabetes and Weight Management: RYGB Group (N=19)
sudden death (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hospitalization for diabetes management (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
coronary bypass graft or stent (Cardiac disorders) | 0 (0) | 2 (8) | 1 (1) | 0 (0)
cardiac arrest - survived (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
presyncope (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
syringomyelia repair (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
bariatric surgery revisions and complications (Surgical and medical procedures) | 8 (11) | 0 (0) | 8 (8) | 0 (0)
Erb's palsy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cancer (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) — 1 prostate (IMWM-band requiring 2 surgical procedures), 1 breast (RYGB)
cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
orthopedic procedures (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) — laminectomy (IMWM-band), hip arthroplasty
renal (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) — surgical repair for urinary incontinence (IMWM-band), acute kidney injury (RYGB), nephrolithiasis (RYGB), urinary tract infection (RYGB)
congestive heart failure hospitalization (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
supraventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
pulmonary embolism (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
psychiatric hospitalizations (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
panniculectomy (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size limits generalizability. Study performed at a single academic medical center. Duration of diabetes and insulin use, as proxies for β-cell function, were not inclusion or exclusion criteria.

Long-term durability of beneficial effects of reducing weight and HbA1c could not be evaluated after 3 years.

Newer bariatric surgical procedures, e.g. sleeve gastrectomy, were not studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No